CLINICAL TRIAL: NCT05267951
Title: Closed-loop Spinal Stimulation for Restoration of Upper Extremity Function After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Chet Moritz, Associate Professor: Division of Physical Therapy, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00013469
Record Dates: First submitted 2021-10-15; First posted 2022-03-07 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Participants who participate in Aim 1 Section of the study will receive open-loop and closed-loop stimulation intervention arms in a randomized order.
  The order of the two interventions in the Aim 2 Section of the study will be the same for all participants enrolled in the Aim 2 Section of the study.
Who Masked: Outcomes Assessor
Masking Description: Functional measurements and all other assessments will be done by an examiner who does not know the order of the intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Open-loop Stimulation (Experimental): Continuous stimulation
  Interventions: Device: Open-loop Stimulation; Other: Functional Task Practice
- Close-loop Stimulation (Experimental): Intended movement-based stimulation.
  Interventions: Device: Close-loop Stimulation; Other: Functional Task Practice

INTERVENTIONS:
Device: Open-loop Stimulation — Spinal cord stimulation will be applied continuously over the skin throughout the intervention session.
  Arms: Open-loop Stimulation
Device: Close-loop Stimulation — Spinal cord stimulation will start and stop based on the signals that come from the sensors placed on upper limb muscle surfaces.
  Arms: Close-loop Stimulation
Other: Functional Task Practice — Exercise therapy consists of repeated functional hand and arm movements
  Other Names: Intensive exercise therapy

SUMMARY:
The purpose of this study is to assess the efficacy of non-invasive (transcutaneous) closed-loop electrical spinal cord stimulation for recovery of upper limb function (Aim 1) and spasticity (Aim 2) following spinal cord injury.

DETAILED DESCRIPTION:
After being informed about the purpose, study timeline, and procedures, all participants giving written informed consent will undergo repeated baseline measurements throughout four weeks, followed by intensive exercise therapy for six weeks.

Next, participants will receive (1) closed-loop stimulation and (2) open-loop stimulation treatment for Aim 1 Section of the study. Stimulation will be delivered non-invasively using skin electrodes on the back of the neck. Each treatment arm will last six weeks. The investigators will determine the order of the treatment arms randomly. For closed-loop stimulation, The investigators will place a sensor on the arm muscles over the skin. This sensor will detect the movement and start the stimulation accordingly.

For Aim 2 Section, intervention arms will consist of (1) transcutaneous stimulation, followed by (2) spasticity-reducing stimulation treatment arms.

There will be a 6-week waiting period between two stimulation arms where participants will not receive any stimulation or exercise therapy. Treatments will last 90 minutes per session, three sessions per week. Overall participation in the study will last ten months: Four weeks baseline + three treatment periods (each will last six weeks) + six weeks waiting period between stimulation treatments + 12 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. has cervical (C8 or higher), incomplete (American Spinal Cord Injury Impairment Scale - C or D) traumatic spinal cord injury, minimum 1-year post-injury
2. has difficulty with hand functions in activities of daily living (e.g., dressing, grooming, feeding)
3. stable medical condition without cardiopulmonary disease or autonomic dysreflexia that would contraindicate participation in upper extremity rehabilitation or testing activities
4. capable of performing simple cued motor tasks
5. has ability to attend intervention/functional task training and assessment sessions 3 times/week
6. has adequate social support to participate in all intervention and baseline/follow-up assessment sessions throughout 40 weeks.
7. has ability to read and speak English

Exclusion Criteria:

1. dependent on ventilation support
2. has implanted stimulator (e.g., pacemaker, vagus nerve stimulator, cochlear implant, etc.) or baclofen pump
3. has metallic devices and implants in the head (e.g., deep brain stimulators, aneurysm clips/coils, and stents, vagus nerve stimulators)
4. has a history or current signs/symptoms of syringomyelia (progressive pain, muscle weakness, and/or sensory loss; deterioration of bowel/bladder function)
5. has autoimmune etiology of spinal cord dysfunction/injury
6. has received botulinum toxin injections in upper extremity muscles in the prior 6 months
7. has tendon transfer or nerve transfer surgery in the upper extremity,
8. taking tizanidine, dantrolene or diazepam
9. has history of seizures or increased risk for seizures
10. has history of chronic headaches or migraines
11. has history of neurologic diseases, such as stroke, multiple sclerosis, traumatic brain injury, etc.
12. has peripheral neuropathy (diabetic polyneuropathy, entrapment neuropathy, etc.)
13. has rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.)
14. has significant medical disease; including uncontrolled systemic hypertension with values above 170/100 mmHg; cardiac or pulmonary disease; uncorrected coagulation abnormalities or need for therapeutic anticoagulation
15. has cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention
16. unhealed fracture, contracture, pressure sore, or frequent urinary tract infections or other illnesses that might interfere with upper extremity rehabilitation or testing activities
17. has a history of severe allergy (i.e., allergic reaction that could not be treated with antihistaminic medication
18. has alcohol and/or drug abuse (subject's verbal statement)
19. has cancer
20. pregnant (Childbearing potential will be asked at screening, baseline, and every subsequent visit in which the subject would receive transcutaneous spinal cord stimulation and/or Transcranial Magnetic Stimulation whether the participant could be pregnant. Pregnancy will be ruled out by an over-the-counter urine pregnancy test for all females of childbearing potential (1) at the time of enrollment, (2) prior to all sessions that include Transcranial Magnetic Stimulation, and also prior to the intervention phases of (3) closed-loop or (4) open-loop stimulation. Additional pregnancy tests may be performed if there is a concern of pregnancy.)
21. lack of ability to fully comprehend, cooperate and/or safely perform study procedures in the investigator's opinion/judgment
22. unable to read and/or comprehend the consent form

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline- Graded Redefined Assessment of Strength, Sensation, and Prehension version 2 | "Repeated measurements once every two weeks throughout the study, an average of 10 months".
  Measurement of upper limb strength, sensation, qualitative prehension, and quantitative prehension (range 0-188, higher score mean better outcome)
Change from baseline- Capabilities of Upper Extremity Test | "Repeated measurements once every two weeks throughout the study, an average of 10 months".
  Measures unilateral and bilateral hand and arm function (range 0-128, higher score mean better outcome)
Change from baseline- Grip and Pinch Force | "Repeated measurements once every two weeks throughout the study, an average of 10 months".
  Grip and pinch force measurement using a dynamometer (higher score mean better outcome)
Change from baseline- Modified Ashworth Scale | "Repeated measurements once every two weeks throughout the study, an average of 10 months".
  Clinician administered assessment of spasticity (range 0-4, lower score mean better outcome)

SECONDARY OUTCOMES:
Change from baseline- International Standards for Neurologic Classification of Spinal Cord Injury - Motor Score | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Standard manual muscle strength examination (Range 0-100 points, higher score mean better outcome)
Change from baseline- International Standards for Neurologic Classification of Spinal Cord Injury - Sensory Score | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Standard examination of dermatomal sensation (range 0-224 points, higher score mean better outcome)
Change from baseline- International Standards of Autonomic Functions after Spinal Cord Injury | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Clinician assessment to document remaining autonomic functions after spinal cord injury
Change from baseline- H-Reflex | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Electrophysiologic measurement of H-reflex (lower Hmax/Mmax ratio mean better outcome)
Change from baseline- Somatosensory Evoked Potentials | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Electrophysiologic evaluation of sensory pathways between the brain and the limb (shorter latency mean better outcome)
Change from baseline- Motor Evoked Potentials | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Electrophysiologic evaluation of motor pathways between the brain and the muscles (higher amplitude mean better outcome)
Change from baseline Spinal Cord Independence Measure Self Report | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Quantification of the level of independence in daily activities (range 0-100 points, higher score mean better outcome)

OTHER OUTCOMES:
Change from baseline- World Health Organization Quality of Life Questionnaire | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Self-reported questionnaire on quality of life (range 0-100 points, higher score mean better outcome)
Change from baseline- Spinal Cord Injury - Functional Index Short-Form | "Baseline"/"At the end of each treatment arm"/"Through study completion"
  Patient-reported questionnaire (range 0-100 points, higher score mean better outcome)
Change from baseline- International Spinal Cord Injury Bowel Function Basic Data Set.v.2.1 | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Patient-reported questionnaire (range 0-47 points, lower score mean better outcome)
Change from baseline- Patient Reported Impact of Spasticity Measure | "Repeated measurements once every eight weeks throughout the study, an average of 10 months".
  Patient-reported questionnaire (range 0-164 points, lower score mean better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Chet Moritz, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inanici F, Samejima S, Gad P, Edgerton VR, Hofstetter CP, Moritz CT. Transcutaneous Electrical Spinal Stimulation Promotes Long-Term Recovery of Upper Extremity Function in Chronic Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1272-1278. doi: 10.1109/TNSRE.2018.2834339. PMID 29877852
- [Background] Inanici F, Brighton LN, Samejima S, Hofstetter CP, Moritz CT. Transcutaneous Spinal Cord Stimulation Restores Hand and Arm Function After Spinal Cord Injury. IEEE Trans Neural Syst Rehabil Eng. 2021;29:310-319. doi: 10.1109/TNSRE.2021.3049133. Epub 2021 Mar 2. PMID 33400652
- [Background] McPherson JG, Miller RR, Perlmutter SI. Targeted, activity-dependent spinal stimulation produces long-lasting motor recovery in chronic cervical spinal cord injury. Proc Natl Acad Sci U S A. 2015 Sep 29;112(39):12193-8. doi: 10.1073/pnas.1505383112. Epub 2015 Sep 14. PMID 26371306